CLINICAL TRIAL: NCT05205668
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of F-652 in Subjects With COVID-19 Pneumonia
Brief Title: Study of F-652 in Subjects With Corona Virus Disease 2019 (COVID-19) Pneumonia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Compound development plan changed
Sponsor: EVIVE Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: EV-652-011
Record Dates: First submitted 2022-01-17; First posted 2022-01-25 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — eflepedocokin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- F-652 Dosage Level 1 (Experimental): IL-22 fusion protein administered intravenously
  Interventions: Biological: F-652
- Placebo (Placebo Comparator): Placebo administered intravenously
  Interventions: Biological: Placebo
- F-652 Dosage Level 2 (Experimental): IL-22 fusion protein administered intravenously
  Interventions: Biological: F-652

INTERVENTIONS:
Biological: F-652 — IL-22 fusion protein administered intravenously
  Arms: F-652 Dosage Level 1; F-652 Dosage Level 2
Biological: Placebo — Placebo administered intravenously
  Arms: Placebo

SUMMARY:
This is a phase 2a, multicenter, randomized, double-blinded, placebo controlled, dose escalation study in adult subjects with COVID-19 pneumonia. The primary objective of this study is to evaluate the overall safety of F-652 in COVID subjects in order to identify safe dose(s) for future studies with adequate patient numbers to demonstrate clinical efficacy.

DETAILED DESCRIPTION:
The study is planned to include 2 cohorts, with enrolled patients being randomized 2:1 in a blinded manner on Day 1, following screening, to F-652 or placebo as follows:

* Cohort 1: subjects will receive up to two intravenous (IV) infusions of F-652 at dose 1 or placebo. Upon completion of Cohort 1, the data monitoring committee (DMC) will convene and review all available safety data to determine if the study can proceed to the next dose level.
* Cohort 2: subjects will receive up to two IV infusions of F-652 at dose 2 or placebo.

Approximately 60 eligible subjects will be enrolled in the study with 30 subjects per dose cohort. Each cohort will have about 20 subjects treated with F-652 and 10 subjects treated with matching placebo.

All randomized subjects will receive standard-of-care treatments for COVID-19 per individual institution standards. Treatment will begin on Day 1 following randomization. Subjects will receive up to two IV infusions of F-652 or matching placebo.

ELIGIBILITY:
Inclusion Criteria: Subjects who meet all of the following criteria will be eligible to participate in the study

* Hospitalized subjects with a positive severe acute respiratory syndrome (SARS)-Corona Virus (CoV)-2 virologic test (nucleic acid amplification test) performed within 2 weeks prior to screening. For subjects with a positive COVID test result within 2 weeks of screening, a confirmatory polymerase chain reaction (PCR) test will be done before randomization.
* Symptoms of moderate illness with COVID-19, which could include any one of the following: fever, cough, sore throat, malaise, headache, muscle pain, nausea, vomiting, diarrhea, loss of taste or smell, shortness of breath with exertion, or respiratory distress.
* Clinical signs suggestive of moderate to severe illness with COVID-19, which could include any one of the following symptoms: respiratory rate ≥ 20 breaths per minutes, heart rate ≥ 90 beats per minute, abnormal saturation of peripheral oxygen (SpO2) defined by pulse oximeter <95% room air at sea level, or lung infiltration on chest X-ray imaging.
* Willingness to provide informed consent and being able to comply with the protocol therapy required monitoring and follow-up.
* Age ≥18 years old.
* Females of childbearing potential (FCBP) must have a negative serum pregnancy test at screening. FCBP and males of reproductive potential must be willing to completely abstain or agree to use a highly effective method of contraception (i.e., less than 1% failure rate) from the time of signing the informed consent and for the duration of study and at least 2 months following the last dose of study drug.

Exclusion Criteria: Subjects who meet any of the following criteria will be excluded from participation in the study:

* Respiratory failure defined based on resource utilization requiring at least one of the following: endotracheal intubation and mechanical ventilation, oxygen delivered by high flow nasal cannula (>40 Liters per minute with fraction of delivered oxygen >0.5), noninvasive positive pressure ventilation, extracorporeal membrane oxygenation (ECMO), or clinical diagnosis of respiratory failure (ie, clinical need for one of the preceding therapies, but preceding therapies unavailable due to resource limitation).
* Septic shock defined by systolic blood pressure < 90 mm Hg, or diastolic blood pressure < 60 mm Hg, or requiring vasopressor use.
* Multi-organ dysfunction or failure based on investigator's determination including sequential organ failure assessment (SOFA) score.
* Unlikely to survive beyond 2 days at the discretion of Investigator.
* Has received high-dose corticosteroids (dexamethasone >12 mg/day or equivalent) for longer than 2 days within 72 hours prior to screening. However, corticosteroids at doses used as standard-of-care treatment for COVID-19 per individual institution standard will be allowed.
* Chronic obstructive pulmonary disease or bronchial asthma requiring treatment within 3 months prior to screening.
* Clinical evidence of active or unstable cardiovascular diseases (i.e. heart failure or acute myocardial infarction) as determined by investigator assessment.
* Active liver disease or hepatic insufficiency or alanine aminotransferase or aspartate aminotransferase level >5 times the upper limit of normal range at screening.
* Severe renal insufficiency requiring dialysis at screening.
* Any of the following abnormal laboratory values: absolute neutrophil count (ANC) < 1,000 per mm3, or platelets count <50,000 per mm3 detected within 48 hours at screening per local lab.
* A history of an invasive malignancy within the past 5 years except for the following circumstances: malignant tumors cured with no recurrence in the past 5 years, completely resected basal cell or squamous cell carcinoma of the skin, and/or completely resected carcinoma in situ of any type.
* Active tuberculosis (TB) or uncontrolled TB, or severe infection caused by bacteria or fungi within 4 weeks prior to screening
* History of human immunodeficiency virus (HIV) infection or hepatitis B or hepatitis C.
* Has received any other investigational therapeutic products within 8 weeks or 5 half-lives, whichever is longer, prior to screening.
* A known serious allergic reaction or hypersensitivity to components of F-652.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with any treatment-emergent adverse events (TEAEs) during the study | Day 1 to Day 60/End of Study (EOS)

SECONDARY OUTCOMES:
Proportion (%) of subjects with any serious adverse events (SAEs) and drug-related adverse events (AEs) during the study | Day 1 to Day 60/EOS
Proportion (%) of subjects with clinically significant abnormality in clinical laboratory tests and ECG during the study | Day 1 to Day 28
Change in parameters for coagulopathy including D-dimer, fibrinogen, coagulation tests and platelet count during the study | Day 1 to Day 28
Change in parameters of cardiac function including N-terminal-pro hormone brain natriuretic peptide (NT-proBNP) or brain natriuretic peptide (BNP) and high-sensitivity cardiac troponin (or troponin) during the study | Day 1 to Day 28
Serum concentration of F-652 at specified timepoints | At predefined timepoints from Day 1 to Day 14/End of Treatment (EOT)
Number of days with oxygen use during the treatment period | Day 1 to Day 14/EOT
Change in the World Health Organization (WHO) 10-point ordinal scale during the study period | Day 1 to Day 14/EOT and Day 28
  The World Health Organization 10-point ordinal scale is developed by a special committee at WHO to measure illness severity over time. The minimum value is 0, the maximum value is 10. Severity increases as the score increases. A 2-point reduction on the score is considered as clinical improvement.
Number of days hospitalized during the treatment period | Day 1 to Day 14/EOT
Proportion (%) of subjects alive and free of respiratory failure during the study period | Day 1 to Day 14/EOT, Day 28, and Day 60/EOS
All-cause mortality rate during the study period | Day 1 to Day 14/EOT, Day 28, and Day 60/EOS

OTHER OUTCOMES:
Exploratory Endpoints - biomarkers | Day 1 to Day 14/EOT
  Changes in biomarkers mainly indicative of lung injury and inflammation

IPD SHARING:
Plan to Share IPD: No